CLINICAL TRIAL: NCT03267563
Title: Implementing to Sustain: Determining the Minimum Necessary Intervention to Maintain a Postpartum Depression Prevention Program (ROSE) in Clinics Providing Prenatal Services to Low-income Women
Brief Title: Minimum Intervention to Maintain a Postpartum Depression Prevention Program in Clinics Serving Low-income Women
Acronym: ROSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Butler Hospital (Other); Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other); Palo Alto Veterans Institute for Research (Other); University of Rochester (Other); University of Massachusetts, Worcester (Other); Pacific Institute for Research and Evaluation (Other)
Responsible Party: Principal Investigator, Jennifer E. Johnson, C. S. Mott Endowed Professor of Public Health, Professor of OBGYN, Professor of Psychiatry and Behavioral Medicine, Michigan State University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: MichiganSUROSE
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Depression, Postpartum
Keywords: prevention; implementation; sustainment; perinatal; pregnancy; postpartum
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Sequential, multiple assignment, randomized trial (SMART) design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced implementation as usual (EIAU) (Experimental): All clinics will receive enhanced implementation as usual (EIAU) that is initial clinical and operational training + tools for sustainment. This occurs once at the beginning of the trial.
  Interventions: Behavioral: EIAU
- Low-intensity coaching and feedback (Experimental): Clinics will receive enhanced implementation as usual (EIAU) plus low-intensity (every 3 months) implementation coaching and feedback (LICF). LICF consists of quarterly clinical and operational coaching and feedback calls, as well as quarterly participation in an implementation collaborative board.
  Interventions: Behavioral: EIAU; Behavioral: LICF
- High-intensity coaching and feedback (Experimental): Clinics will receive enhanced implementation as usual (EIAU) plus high-intensity (every month) implementation coaching and feedback (HICF). HICF consists of monthly clinical and operational coaching and feedback calls, monthly participation in an implementation collaborative board, and on call technical assistance.
  Interventions: Behavioral: EIAU; Behavioral: LICF; Behavioral: HICF

INTERVENTIONS:
Behavioral: EIAU — Enhanced implementation as usual consists of initial training and problem-solving plus planning for sustainment,
Behavioral: LICF — Enhanced implementation plus low intensity will have received initial training and problem-solving plus planning for sustainment and after that every 3 months will receive one clinical and one operational telephone "booster" meeting.
  Arms: High-intensity coaching and feedback; Low-intensity coaching and feedback
Behavioral: HICF — Enhanced implementation plus high intensity will receive will receive everything that the clinics in LICF receive, but at a higher intensity.
  Arms: High-intensity coaching and feedback

SUMMARY:
Postpartum depression (PPD) is common and can have lasting consequences for mother and child. ROSE is an intervention to prevent PPD, delivered during pregnancy in outpatient prenatal settings. ROSE has been found to significantly reduce cases of PPD in multiple randomized trials in community prenatal settings with racially and ethnically diverse low-income pregnant women. Requests for ROSE training and recent policy changes supporting payment for comprehensive perinatal services to underserved populations suggest a context ripe for embedding ROSE in prenatal clinics long-term. Given the need for return on investment studies about sustainment efforts, we propose a Sequential Multiple Assignment Randomized (SMART) Trial of the effectiveness and cost-effectiveness of a stepwise approach to sustainment of ROSE in 90 outpatient clinics providing prenatal care to pregnant women on public assistance in 6 U.S. states. In Year 1, all clinics will receive enhanced implementation as usual (EIAU; initial training + tools for sustainment). At the first time at which a clinic is determined to be at risk for failure to sustain (i.e., at 3, 6, 9, 12, 15 months), that clinic will be randomized to receive either: (1) no additional implementation support (i.e., EIAU only), or (2) low-intensity coaching and feedback (LICF). If clinics receiving LICF are still found to be at risk at subsequent assessments, they will be randomized to either (1) EIAU + LICF only, or (2) high-intensity coaching and feedback (HICF). Additional study follow-up interviews will occur at 18, 24, and 30 months, but no implementation intervention will occur after 18 months. Outcomes include: 1. Sustainment of core program elements at each time point and total length of time ROSE services were provided and were provided with at least moderate fidelity. 2. Health impact (PPD rates over time at each clinic) and reach. 3. ROI (costs, cost-offsets, and cost-effectiveness) of each sustainment step. Hypothesized mechanisms include sustainment of clinical and organizational capacity to deliver core elements, and engagement/ownership. The study will also examine predictors, tailoring variables, and implementation processes to determine which kinds of clinics need which level of sustainment support and when. To our knowledge, this study will be the first randomized trial evaluating the ROI of a stepped approach to sustainment, a critical unanswered question in implementation science.

DETAILED DESCRIPTION:
A recent expert consensus report concluded that, "Little is known about how well or under what conditions health innovations are sustained and their gains maintained once they are put into practice. Implementation science typically focuses on uptake by early adopters. The later-stage challenges of sustaining evidence-supported interventions receive too little attention." This report placed high priority on conducting return on investment (ROI) studies to determine how much is gained when effective programs are sustained, and cost-benefit trade-offs for effort required to sustain.1 Information is especially needed for preventive behavioral health interventions for adults in outpatient medical (e.g., primary care; OBGYN) settings.

Postpartum depression (PPD) is common and can have serious and lasting consequences for mother and child, including maternal increased risk for suicide, compromised functional status, and adverse infant developmental outcomes. Prevalence of PPD is ~13% in the 12 weeks after childbirth, with rates up to 50% among low-income women, who are especially vulnerable to the consequences of PPD. Outpatient clinics offering prenatal care are an opportune place to deliver PPD prevention services because most women will visit while pregnant. Recent guidelines suggest that prenatal clinics should screen for PPD after birth and refer once it is identified. Unfortunately, prenatal clinics do not routinely do anything to prevent PPD from occurring.

The ROSE Program (Reach Out, Stay Strong, Essentials for mothers of newborns) is a small-group intervention to prevent PPD that is delivered during pregnancy in outpatient prenatal settings. ROSE is the only PPD preventative intervention that (1) has been found to significantly reduce cases of PPD in multiple randomized trials, and (2) has been tested in community prenatal settings with racially and ethnically diverse low income pregnant women. ROSE consists of four 90-minute group sessions and a 50-minute individual booster session after delivery. Requests for ROSE training in Philadelphia and nationwide in Japan, and recent policy changes supporting payment for comprehensive perinatal services (including behavioral health care) to underserved populations all suggest a context ripe for embedding ROSE in prenatal clinics long-term. Given the need for ROI studies about sustainment efforts and that ROSE is well-positioned for implementation and sustainment research, we propose a Sequential Multiple Assignment Randomized (SMART) Trial of the effectiveness and cost-effectiveness of a stepwise approach to sustainment of ROSE in 90 outpatient clinics providing prenatal care to pregnant women on public assistance accross the US. Our conceptual framework comes from RE-AIM and a review on sustainment by Co-I Wiltsey-Stirman,3 with sustainment strategies based on the Replicating Effective Programs (REP) framework. All clinics will receive enhanced implementation as usual (EIAU; initial training + tools for sustainment). Clinics will be assessed using surveys and qualitative interviews 9 times over 2.5 years after receiving EIAU. Clinics at risk for failure to sustain operationally (defined as no ROSE intervention in 3 months and none planned) and/or clinically (defined as low fidelity to ROSE core elements) will be randomized to receive additional sustainment support for up to 18 months after baseline. At the first time period at which a clinic is determined to be at risk (i.e., at 3, 6, 9, 12, or 15 months), that clinic will be randomized to receive either: (1) no additional implementation support (EIAU only), or (2) EIAU plus low-intensity (every 3 months) coaching and feedback (LICF). If clinics receiving LICF are still at risk at subsequent monitoring periods, they will be randomized to (1) EIAU + LICF only, or (2) EIAU + LICF + high-intensity (monthly) coaching and feedback (HICF). Additional study follow-up interviews will occur at 18, 24, and 30 months, but no implementation intervention will occur after 18 months. We will assess costs and benefits of sustainment strategies. Aims are to:

Compare effectiveness of each sustainment step for the following final and proximal OUTCOMES:

1. Sustainment of core program elements at each time point, and total length of time in weeks that: (i) any ROSE services were provided, and (ii) were provided with adequate fidelity to core elements (primary).
2. Health impact (e.g., PPD rates over time at each clinic) and reach (number of patients enrolled in and completing the ROSE program).
3. Return on Investment (costs and cost-effectiveness of each sustainment step).
4. Hypothesized mechanisms include sustainment of: (a) clinical and organizational capacity to deliver core elements, and (b) a sense of engagement/ownership by key clinic staff, Examine predictors and processes to determine which kinds of clinics need which level of support.
5. Explore which clinic characteristics (e.g., organizational and state policy contexts) and hypothesized mechanisms (Aim 4) are associated with best sustainment to determine tailoring variables for choosing/sequencing EIAU, LICF, HICF in the future.
6. Document implementation/sustainment effort processes, their timing relative to desired outcomes, critical incidents to explore factors most related to sustainment after accounting for hypothesized mechanisms.

To our knowledge, this study will be the first randomized trial evaluating the ROI of a stepped approach to sustainment, a critical unanswered question in implementation science. The study will also examine a set of strategies to promote sustainment of an effective PPD prevention intervention for low-income women, reducing negative consequences for mother and child. The proposal directly addresses the goal of PAR-16-238 to conduct longitudinal studies on "factors that contribute to the sustainability of evidence-based interventions," to test strategies to improve quality of care among underserved populations, examine mediators and moderators, and examine cost-effectiveness or other economic outcomes. Thus, the study will advance implementation science, knowledge of implementation science mechanisms, and clinical care for an at-risk population.

ELIGIBILITY:
Study enrollment and randomization takes place at the clinic level. Study participants will be clinical and operational staff representatives of participating clinics.

To be included in the study, clinics will:

* provide outpatient prenatal services
* estimate that at least 50% of their pregnant patients receive some kind of public assistance (such as federal or state assistance in the form of cash assistance such as Temporary Assistance for Needy Families [TANF], food stamps, subsidized housing, and/or health care such as Medicaid)
* have at least 10 new pregnant women per month on average (i.e., enough patient flow to run ROSE)
* agree to study procedures.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 791 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Sustainment of core program elements | Measured at 3, 6, 9, 12, 15, 18, 24, and 30 months after baseline
  The total length of time that ROSE services were provided with adequate (75% or more) fidelity to core elements. The ROSE Session-by-Session Adherence Scale, a self-rated intervention fidelity scale completed by ROSE interventionists after each session. The outcome for each time point (i.e., quarter) will be the mean % of core elements delivered that should have been delivered at each ROSE session (mean [# of core elements delivered/# core elements should have been delivered] at each session; zero if no sessions were completed).

SECONDARY OUTCOMES:
Total length of time any ROSE services were offered | Measured at 3, 6, 9, 12, 15, 18, 24, and 30 months after baseline
  The total length of time any ROSE services were provided will be tracked using a monthly calendar method
Health impact: Postpartum depression (PPD) rates over time at each clinic | Quarterly over 30 months
  Quarterly, we will ask each clinic to report the following overall numbers: (1) # of women who should have come for their 6-week postpartum appointment; (2) # who came; (3) # that were screened for PPD; (4) # who screened positive for PPD. We will also collect this information for 4 quarters (12 months) prior to baseline. We will use these numbers to calculate PPD rates for each time period. Although though not every woman in the clinic will receive ROSE, we chose to track overall PPD rates at each clinic because: (1) the study examines larger-scale sustainment aimed at clinic-wide (and eventually population-wide) outcomes; and (2) the clinic-level outcomes are primary; not consenting individual patients makes the needed sample size (90 clinics) feasible.
ROSE Intervention reach | Quarterly over 30 months
  # patients receiving ROSE and # of patients who complete at least 3 of 5 sessions
Cost-effectiveness | Measured at 3, 6, 9, 12, 15, 18, 24, and 30 months after baseline
  We will analyze 4 cost-effectiveness (CE) outcome measures: (1) a primary clinical outcome, number of PPD cases averted, estimated as the change in PPD rate at the clinic (post-pre)*(clinic's caseload), (2) another clinical outcome, number of quality-adjusted life years (QALYs) saved, computed from the primary outcome using Morrell et al.'s model, (3) an implementation process outcome, number of clients served with fidelity, and (4) a sustainment outcome, months of additional service delivery. The latter 2 measures have little measurement error.

OTHER OUTCOMES:
Hypothesized mechanism: Sustainment of clinical and organizational capacity to deliver core elements | Measured at baseline, 3, 6, 9, 12, 15, 18, 24, and 30 months after baseline
  Organizational Capacity subscale of the Program Assessment Sustainability Tool (PSAT). Secondary measures of this construct include number of people trained who have time to deliver ROSE and clinic's ability to manage space, scheduling, and reimbursement for ROSE
Hypothesized mechanism: Sustainment of a sense of engagement/ownership by key clinic staff. | Measured at baseline, 3, 6, 9, 12, 15, 18, 24, and 30 months after baseline
  The sum of 4 PSAT subscales: Political Support, Partnerships, Communications, and Strategic Planning. The Staff section of the NHS's Sustainability Model and Guide and investment in addressing PPD will be secondary measures

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Johnson, Ph.D., Principal Investigator — Michigan State University; Raven Miller, M.A., Study Director — Michigan State University
Locations (1):
- Michigan State University, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
After data have been collected and study results published, de-identified data will be made available to other qualified researchers upon request, on a CD or other electronic means compatible with our systems. The request will be evaluated by the PIs to ensure that it meets reasonable standards of scientific integrity.
  We have use standard measures where possible in order to promote data sharing and integration into larger databases and to allow other researchers to analyze the data, including conducting meta-analyses. We will work on the data dictionary throughout the study. Data checking will occur regularly. We will submit primary results for publication by the end of the project period, and will have final de-identified datasets and data dictionaries available by CD within the required time frame.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the main results
Access Criteria: De-identified data will be made available for scientific inquiry

REFERENCES:
- [Derived] Johnson JE, Wiltsey-Stirman S, Sikorskii A, Miller T, Poleshuck E, Simas TAM, Carravallah L, Miller R, Zlotnick C. Outcomes of the ROSE Sustainment (ROSES) Study, a sequential multiple assignment randomized implementation trial to determine the minimum necessary intervention to sustain a postpartum depression prevention program in agencies serving low-income pregnant people. Implement Sci. 2025 Feb 10;20(1):9. doi: 10.1186/s13012-025-01420-z. PMID 39930503
- [Derived] Johnson JE, Wiltsey-Stirman S, Sikorskii A, Miller T, King A, Blume JL, Pham X, Moore Simas TA, Poleshuck E, Weinberg R, Zlotnick C. Protocol for the ROSE sustainment (ROSES) study, a sequential multiple assignment randomized trial to determine the minimum necessary intervention to maintain a postpartum depression prevention program in prenatal clinics serving low-income women. Implement Sci. 2018 Aug 22;13(1):115. doi: 10.1186/s13012-018-0807-9. PMID 30134941